CLINICAL TRIAL: NCT04729647
Title: Immature Granulocyte Count and Delta Neutrophil Index as New Predictive Factors for Axillary Metastasis of Breast Cancer
Brief Title: Immature Granulocyte Count and Delta Neutrophil Index Factors for Axillary Metastasis of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Mehmet Buğra Bozan, Professor, Assistant, Kahramanmaras Sutcu Imam University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19
Record Dates: First submitted 2021-01-01; First posted 2021-01-28 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Breast Cancer Invasive
Keywords: Delta Neutrophil Index; Immature Granulocyte Count; Netrophil Lymphocyte Ratio; Breast Cancer; Axillary Metastasis
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy; Sentinel Lymph Node Biopsy; Blood Cell Count; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: patients without axillary metastases and who did not receive neoadjuvant treatment were examined by dividing them into two groups as pathologically non-metastatic (Group NM) and metastasized (Group M) in axillary lymph node sampling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Axillary Lymph Node Metastasis (Other)
  Interventions: Procedure: Mastectomy

INTERVENTIONS:
Procedure: Mastectomy — Mastectomy for breast cancer Blood sample for Complete Blood Cell Count and other blood parameters (Delta Neutrophil Index, Immature Granulocyte Count)
  Other Names: Sentinel Lymph Node; Axillary dissection; Complete Blood Count; Delta Neutrophil Index; Immature Granulocyte Count; Delta Neutrophil Index and Immature Granulocyte Count; Blood sample for Complete Blood Cell Count

SUMMARY:
Background: Breast cancer ranks first among cancer types seen in women in our country and all over the world, and second after lung cancer in cancer-related deaths. Despite the recent increase in its incidence, mortality has decreased due to early diagnosis and advances in neoadjuvant therapy. Classically, lymph node status, tumor size, histological type and grade, age, and ethnicity are prognostic factors for this type of cancer. Bone marrow activation results from malignancies and inflammation. Tumor-related inflammation has gained importance in each stage of tumorigenesis. Host-dependent systemic inflammatory response has been found to be effective in carcinogenesis, tumor development and progression. Inadequately controlled or uncontrolled inflammatory activity may be responsible for malignant transformation. Inflammatory cell stimulation occurs in lymph node metastasis and distant organ metastases like primary tumor.As the cornerstone of the adaptive immune system, lymphocytes inhibit tumor cell proliferation, migration and destroy metastatic lesions. Monocyte-macrophages inhibit angiogenesis, tumor growth and distant spread. On the other hand, tumor-induced neutrophils can accelerate tumor metastasis. Many studies have examined the relationship between the ratios between different cell types, such as the platelet-lymphocyte ratio (PLR), and the neutrophil-lymphocyte ratio (NLR), with malignant tumors(4,10).Apart from these, mean platelet volume (MPV), which can be automatically studied in routine blood counts and shows platelet activation, has been used to show tumor activity in breast, stomach, colon and ovarian cancers.

Recent studies have identified the delta neutrophil index (DNI), which indicates the percentage of immature granulocytes (IG) in peripheral blood due to increased bone marrow activation in inflammatory conditions.It is based on counting granulocyte precursor cells under microscope. With the technological developments,IG count and DNI can be automatically evaluated from complete blood count parameters in automated systems.

In this study,the investigators aimed to determine the diagnostic value of preoperative IG number and DNI level before clinical detection of axillary lymph node metastasis, which plays an important role in the prognosis of breast cancer, and to compare these parameters with other routine inflammation markers such as white blood cell count (WBC), MPV, NLR and PLR.

Material - Methods:Patients who were older than eighteen and operated for breast pathology in Kahramanmaras Sutcu Imam University,Department of General Surgery between February 2015 and February 2020 were evaluated retrospectively.Patient data were obtained from patient epicrisis forms and preoperative laboratory and postoperative pathology results recorded in the computer system.Demographic data of the patients,routine blood tests,preoperative imaging methods, preoperative tumor size,presence of axillary lymph node metastasis and distant organ metastasis,presence of pathological axillary lymph node metastasis in the postoperative period were evaluated.

In the preoperative period, patients without axillary metastases and who did not receive neoadjuvant treatment were examined by dividing them into two groups as pathologically non-metastatic(Group NM) and metastasized(Group M) in axillary lymph node sampling.

White blood cell(WBC)count,neutrophil count,lymphocyte count,platelet count,mean platelet volume(MPV),IG count and DNI(IG percentage)were measured using an automated hematological analyzer from blood samples obtained at the preoperative previous month of surgery.Neutrophil to lymhpocyte ratio(NLR) and platelet to lymphocyte ratio(PLR) were manually calculated from the complete blood cell results.

DETAILED DESCRIPTION:
Background: Breast cancer ranks first among cancer types seen in women in our country and all over the world, and second after lung cancer in cancer-related deaths. Despite the recent increase in its incidence, mortality has decreased due to early diagnosis and advances in neoadjuvant therapy. Classically, lymph node status, tumor size, histological type and grade, age, and ethnicity are prognostic factors for this type of cancer. Bone marrow activation results from malignancies and inflammation. Tumor-related inflammation has gained importance in each stage of tumorigenesis. Host-dependent systemic inflammatory response has been found to be effective in carcinogenesis, tumor development and progression. Inadequately controlled or uncontrolled inflammatory activity may be responsible for malignant transformation. Inflammatory cell stimulation occurs in lymph node metastasis and distant organ metastases like primary tumor.As the cornerstone of the adaptive immune system, lymphocytes inhibit tumor cell proliferation, migration and destroy metastatic lesions. Monocyte-macrophages inhibit angiogenesis, tumor growth and distant spread. On the other hand, tumor-induced neutrophils can accelerate tumor metastasis. Many studies have examined the relationship between the ratios between different cell types, such as the platelet-lymphocyte ratio (PLR), and the neutrophil-lymphocyte ratio (NLR), with malignant tumors.Apart from these, mean platelet volume (MPV), which can be automatically studied in routine blood counts and shows platelet activation, has been used to show tumor activity in breast, stomach, colon and ovarian cancers.

Recent studies have identified the delta neutrophil index (DNI), which indicates the percentage of immature granulocytes (IG) in peripheral blood due to increased bone marrow activation in inflammatory conditions.It is based on counting granulocyte precursor cells under microscope. With the technological developments,IG count and DNI can be automatically evaluated from complete blood count parameters in automated systems.

In this study, investigators aimed to determine the diagnostic value of preoperative IG number and DNI level before clinical detection of axillary lymph node metastasis, which plays an important role in the prognosis of breast cancer, and to compare these parameters with other routine inflammation markers such as white blood cell count (WBC), MPV, NLR and PLR.

Material - Methods:Patients who were older than eighteen and operated for breast pathology in Kahramanmaras Sutcu Imam University,Department of General Surgery between February 2015 and February 2020 were evaluated retrospectively.Patient data were obtained from patient epicrisis forms and preoperative laboratory and postoperative pathology results recorded in the computer system.Demographic data of the patients,routine blood tests,preoperative imaging methods, preoperative tumor size,presence of axillary lymph node metastasis and distant organ metastasis,presence of pathological axillary lymph node metastasis in the postoperative period were evaluated.

In the preoperative period, patients without axillary metastases and who did not receive neoadjuvant treatment were examined by dividing them into two groups as pathologically non-metastatic(Group NM) and metastasized(Group M) in axillary lymph node sampling.

White blood cell(WBC)count,neutrophil count,lymphocyte count,platelet count,mean platelet volume(MPV),IG count and DNI(IG percentage)were measured using an automated hematological analyzer from blood samples obtained at the preoperative previous month of surgery.Neutrophil to lymhpocyte ratio(NLR) and platelet to lymphocyte ratio(PLR) were manually calculated from the complete blood cell results.

Statistical Evaluation:IBM-Statistical Package for Social Sciences (SPSS) version 20 was used for statistical analysis. In the evaluation between independent groups;normal distribution was checked for the kolmogorov-simirnov test.While student t test or Mann Whitney U test was used in the evaluation of numerical data according to the conformity of the data to normal distribution,chi-square test was used in the evaluation of categorical data.Multivariate analysis was performed with parameters found to be significant in the evaluation of univariate analysis and predictive values of preoperative blood parameters were calculated.ROC analysis was performed to evaluate the effectiveness of WBC, NLR, PLR, DNI, IG number and MPV values,and sensitivity,specificity values and cut-off values were obtained. Numerical values are expressed as median(minimum - maximum values), categorical values as percentage (%).

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer (invasive ductal carcinoma, invasive lobular carcinoma, mixed invasive ductal lobular carcinoma, mucinous carcinoma, medullary carcinoma, micropapillary carcinoma)
* Clinically negative axillarry metastasis(without neoadjuvant chemotherapy/radiotherapy)
* Pathologically positive or negative axillary metastasis
* No missing data.

Exclusion Criteria:

* Patients who underwent surgery for benign breast disease (such as fibroadenomas, garnulomatous mastitis, hamartomas)
* Patients with other breast malignancies other than invasive breast carcinoma (ductal carcinoma in situ, fibrosarcomas, neuroendocrine tumors, myofibroblastomas, phyllodes tumors)
* Clinically preoperative positive axillary metastasis
* Preoperative patients with distant organ metastasis
* Patients who received neoadjuvant chemotherapy / radiotherapy in the preoperative period
* Patients with missing data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Determination of preoperative axillary metastasis in clinically negative patients | preoperative period
  DNI and IG count calculated automatically in blood samples of the preoperative period of the invasive breast cancer patients

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koc Z, Saglam Z. Determination of the Knowledge and the Practice of Female Patients about breast cancer, Preventive Measures and Breast Self Examination and Effectiveness of Education. Eur J Breast Heal. 2009;5(1):25-33.
- [Background] Marin Hernandez C, Pinero Madrona A, Gil Vazquez PJ, Galindo Fernandez PJ, Ruiz Merino G, Alonso Romero JL, Parrilla Paricio P. Usefulness of lymphocyte-to-monocyte, neutrophil-to-monocyte and neutrophil-to-lymphocyte ratios as prognostic markers in breast cancer patients treated with neoadjuvant chemotherapy. Clin Transl Oncol. 2018 Apr;20(4):476-483. doi: 10.1007/s12094-017-1732-0. Epub 2017 Aug 7. PMID 28785911
- [Background] DeSantis CE, Ma J, Gaudet MM, Newman LA, Miller KD, Goding Sauer A, Jemal A, Siegel RL. Breast cancer statistics, 2019. CA Cancer J Clin. 2019 Nov;69(6):438-451. doi: 10.3322/caac.21583. Epub 2019 Oct 2. PMID 31577379
- [Background] Peng Y, Chen R, Qu F, Ye Y, Fu Y, Tang Z, Wang Y, Zong B, Yu H, Luo F, Liu S. Low pretreatment lymphocyte/monocyte ratio is associated with the better efficacy of neoadjuvant chemotherapy in breast cancer patients. Cancer Biol Ther. 2020;21(2):189-196. doi: 10.1080/15384047.2019.1680057. Epub 2019 Nov 4. PMID 31684807
- [Background] Miklikova S, Minarik G, Sedlackova T, Plava J, Cihova M, Jurisova S, Kalavska K, Karaba M, Benca J, Smolkova B, Mego M. Inflammation-Based Scores Increase the Prognostic Value of Circulating Tumor Cells in Primary Breast Cancer. Cancers (Basel). 2020 May 1;12(5):1134. doi: 10.3390/cancers12051134. PMID 32369910
- [Background] Elyasinia F, Keramati MR, Ahmadi F, Rezaei S, Ashouri M, Parsaei R, Yaghoubi M, Elyasinia F, Aboutorabi A, Kaviani A. Neutrophil-Lymphocyte Ratio in Different Stages of Breast Cancer. Acta Med Iran. 2017 Apr;55(4):228-232. PMID 28532133
- [Background] Mieog JS, van der Hage JA, van de Velde CJ. Preoperative chemotherapy for women with operable breast cancer. Cochrane Database Syst Rev. 2007 Apr 18;2007(2):CD005002. doi: 10.1002/14651858.CD005002.pub2. PMID 17443564
- [Background] Bozan MB, Yazar FM, Kale IT, Yuzbasioglu MF, Boran OF, Azak Bozan A. Delta Neutrophil Index and Neutrophil-to-Lymphocyte Ratio in the Differentiation of Thyroid Malignancy and Nodular Goiter. World J Surg. 2021 Feb;45(2):507-514. doi: 10.1007/s00268-020-05822-6. Epub 2020 Oct 16. PMID 33067685
- [Background] Singh R, Mishra MK, Aggarwal H. Inflammation, Immunity, and Cancer. Mediators Inflamm. 2017;2017:6027305. doi: 10.1155/2017/6027305. Epub 2017 Nov 6. No abstract available. PMID 29234189
- [Background] Ibrahim A, Serkan YF, Tuba A, Erol B, Lutfi P. Can Neutrophil to Lymphocyte Ratio Be a Predictor Tool for The Non-Sentinel Lymph Node Metastasis in Breast Cancer? Chirurgia (Bucur). 2019 Jan-Feb;114(1):83-88. doi: 10.21614/chirurgia.114.1.83. PMID 30830848
- [Background] Taskaynatan H, Alacacioglu A, Kucukzeybek Y, Varol U, Yildiz Y, Salman T, Oflazoglu U, Tarhan MO. Is Monitoring Mean Platelet Volume Necessary in Breast Cancer Patients? Open Med (Wars). 2018 Oct 4;13:450-455. doi: 10.1515/med-2018-0067. eCollection 2018. PMID 30426082
- [Background] Li MM, Yue CX, Fu S, Zhang X, Zhao CJ, Wang RT. Platelet Volume Is Reduced In Metastasing Breast Cancer: Blood Profiles Reveal Significant Shifts. Cancer Manag Res. 2019 Oct 24;11:9067-9072. doi: 10.2147/CMAR.S221976. eCollection 2019. PMID 31695497
- [Background] Song Y, Yang Y, Gao P, Chen X, Yu D, Xu Y, Zhao J, Wang Z. The preoperative neutrophil to lymphocyte ratio is a superior indicator of prognosis compared with other inflammatory biomarkers in resectable colorectal cancer. BMC Cancer. 2017 Nov 10;17(1):744. doi: 10.1186/s12885-017-3752-0. PMID 29126400
- [Background] Barut O, Demirkol MK, Bilecan EB, Sahinkanat T, Resim S. The Delta Neutrophil Index is an Early Predictive Marker of Acute Pyelonephritis in Patients with Ureteral Stone. J Coll Physicians Surg Pak. 2020 Nov;30(11):1149-1154. doi: 10.29271/jcpsp.2020.11.1149. PMID 33222730
- [Background] De Giorgi U, Mego M, Scarpi E, Giordano A, Giuliano M, Valero V, Alvarez RH, Ueno NT, Cristofanilli M, Reuben JM. Association between circulating tumor cells and peripheral blood monocytes in metastatic breast cancer. Ther Adv Med Oncol. 2019 Aug 14;11:1758835919866065. doi: 10.1177/1758835919866065. eCollection 2019. PMID 31452692